CLINICAL TRIAL: NCT04332211
Title: Pseudoephedrine Prophylaxis for Prevention of Middle Ear Barotrauma in Hyperbaric Oxygen Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Siamak Moayedi, MD, Assistant Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HP-00090947
Record Dates: First submitted 2020-03-28; First posted 2020-04-02 (Actual); Results first posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2024-12

CONDITIONS: Barotrauma;Ear
Keywords: Pseudoephedrine; Hyperbaric oxygen therapy; prophylaxis
MeSH Terms: interventions — Hyperbaric Oxygenation; Pseudoephedrine

STUDY DESIGN:
Intervention Model Description: The study will employ a prospective randomized double-blind placebo control study design (enrollment ratio 1:1) to compare whether pseudoephedrine is more effective than placebo in preventing barotrauma during HBOT
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: prospective randomized double-blind placebo control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Pseudoephedrine Group (Experimental): Patients randomized to pseudoephedrine prior to hyperbaric therapy
  Interventions: Procedure: Hyperbaric Oxygen Therapy; Drug: Pseudoephedrine 60 MG
- Placebo Group (Placebo Comparator): Patients randomized to placebo prior to hyperbaric therapy
  Interventions: Procedure: Hyperbaric Oxygen Therapy; Drug: Placebo oral tablet

INTERVENTIONS:
Procedure: Hyperbaric Oxygen Therapy — Hyperbaric oxygen therapy (HBOT) utilizes 100% oxygen delivery at a pressure greater than 1 atmosphere for the treatment of various emergent medical conditions.
Drug: Pseudoephedrine 60 MG — administer either pseudoephedrine or placebo orally to patients requiring hyperbaric oxygen therapy
  Arms: Pseudoephedrine Group
Drug: Placebo oral tablet — administer either pseudoephedrine or placebo orally to patients requiring hyperbaric oxygen therapy
  Arms: Placebo Group

SUMMARY:
Hyperbaric oxygen therapy (HBOT) utilizes 100% oxygen delivery at a pressure greater than 1 atm for the treatment of various emergent medical conditions including carbon monoxide poisoning. The most commonly associated complication of HBOT is middle ear barotrauma (MEB) which occurs when the eustachian tube does not allow air to enter the middle ear space to equalize the pressure between the ambient environment and the inner ear. Patients experiencing MEB usually feel pressure or pain in their ear(s). The spectrum of symptoms ranges from sensation of ear fullness and muffled hearing to severe pain, vertigo and tympanic membrane rupture. The incidence of MEB, depending on the definition used is between 2-45%. The severe discomfort associated with MEB sometimes causes HBOT to be postponed or abandoned. Last year 27/991 treatments at our Center for Hyperbaric and Dive Medicine were aborted due to MEB. Currently there is no objective criteria for predicting which patients will experience these complications, nor is there consensus on effective prevention measures. At our facility, oxymetazoline, a topical nasal decongestant, is the standard rescue medication administered for patients that have symptoms of MEB during HBOT. This is despite two negative studies showing that this medication does not work any better than placebo. Other studies involving scuba divers and airplane travelers showed that oral pseudoephedrine is effective in decreasing MEB. However, the use of pseudoephedrine for patients undergoing HBOT has not been studied. The investigators plan to perform a randomized double blind placebo control trial to determine if pseudoephedrine is effective in decreasing the rate of MEB during HBOT.

DETAILED DESCRIPTION:
Aim 1: To investigate the efficacy of pre-treatment with oral pseudoephedrine 60mg for decreasing MEB during HBOT.

Hypothesis: Patients randomized to pseudoephedrine will have a lesser need for oxymetazoline rescue therapy while being compressed. They will also report less ear pain once at pressure compared to patients receiving placebo.

Aim 2: To measure the incidence of MEB during HBOT. The investigators will also identify factors (age, gender, medical history) that could predispose an individual to developing MEB during HBOT.

Hypothesis: The incidence of MEB defined as requiring stopping compression of the chamber and oxymetazoline rescue will be greater than 30%. Female sex, age above 60, and prior history of ear conditions will be associated with development of MEB.

ELIGIBILITY:
Inclusion Criteria:

* New patient requiring HBOT (either inpatient or outpatient)
* Age greater than or equal to 18 years and less than 80 years
* Fluent in English
* Full decision capacity
* Able and medically cleared to swallow a pill

Exclusion Criteria:

* Contraindication to pseudoephedrine (MAOI use, pregnancy, glaucoma, heart disease, allergy to drug class)
* SBP >160
* DBP > 90
* HR >100
* Decongestant/antihistamine/pseudoephedrine/nasal steroid/oxymetazoline use within 12 hours.
* Prisoner
* Intubated
* Unable take PO meds

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-07-12 (Actual); Study Completion 2023-07-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Siamak Moayedi, MD, Principal Investigator — University of Maryland School of Medicine, Department of Emergency Medicine
Locations (1):
- University of Maryland Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pseudoephedrine Group | Placebo Group
Started | 40 | 41
Completed | 40 | 41
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: analyzed population were all enrolled subjects who took the study pill within the appropriate time and underwent hyperbaric oxygen therapy.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pseudoephedrine Group | Placebo Group | Total
Number analyzed (Participants) | 40 | 41 | 81
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 40 | 41 | 81
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (15) | 53 (12) | 54.5 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 17 | 27
  Male | 30 | 24 | 54
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 40 | 41 | 81
Region of Enrollment [Number; unit: participants]
  United States | 40 | 41 | 81

OUTCOME MEASURES:

1. Primary Outcome: Requirement of Oxymetalozine Rescue for Ear Pain During Hyperbaric Therapy Compression
Description: middle ear barotrauma will be sensed as pain and inability to "clear" the ear to pressure during chamber pressurization. If the patient requires rescue oxymetazoline nasal spray therapy (usual care) they will be counted as having developed middle ear barotrauma.
Time Frame: 12 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Pseudoephedrine Group | Placebo Group
Number analyzed (Participants) | 40 | 41
Participants | 8 | 11

2. Secondary Outcome: Middle Ear Barotrauma Documentation Based on Otoscopy
Description: visual inspection of the tympanic membrane after completion of hyperbaric oxygen therapy by the attending physician and classification based on the Teed score. We are only measuring no injury versus any injury.
Time Frame: 1 minute
Measure: Count of Participants; unit: Participants
Arm/Group | Pseudoephedrine Group | Placebo Group
Number analyzed (Participants) | 40 | 41
Participants | 6 | 11

3. Secondary Outcome: Patient Description of Ear Pain
Description: Patients will be asked to provide a numerical scale level of pain before and after hyperbaric therapy. The scale is from 0 to 10. We only are interested in no pain versus presence of any pain.
Time Frame: 1 minute
Measure: Count of Participants; unit: Participants
Arm/Group | Pseudoephedrine Group | Placebo Group
Number analyzed (Participants) | 40 | 41
Participants | 5 | 12

ADVERSE EVENTS:
Time Frame: 4 hours
Description: no adverse events were expected and none occurred
Arm/Group | Pseudoephedrine Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/41
Other Adverse Events (participants affected / at risk) | 0/40 | 0/41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-01-17): https://cdn.clinicaltrials.gov/large-docs/11/NCT04332211/Prot_SAP_002.pdf
  • Informed Consent Form (2023-03-30): https://cdn.clinicaltrials.gov/large-docs/11/NCT04332211/ICF_003.pdf